CLINICAL TRIAL: NCT03183700
Title: The Value of HPV DNA Testing Using Self-collected Sampling in Non Attendees Cervical Cancer Screening and Molecular Triage Strategies on Self-sampled Material for HPV Positive Women.
Brief Title: Self Collected Sampling in Non-attendees Cervical Cancer Screening: DNA Test and Molecular Triage for HPV Positive Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Prevention and Research Institute, Italy (Other)
Collaborators: Istituto Toscano Tumori (Other)
Responsible Party: Principal Investigator, Francesca Carozzi, Biologist Director, Cancer Prevention and Research Institute, Italy
Allocation: Randomized | Model: Parallel | Purpose: Screening
Other Study IDs: F121I14000310002
Record Dates: First submitted 2017-05-16; First posted 2017-06-12 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Cervical Cancer
Keywords: Screening HPV; Self sampling; DNA Methylation
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control arm 1 (Other): The women will receive the usual recall with a new invitation letter with a prefixed appointment.
  Interventions: Other: Cervical ThinPrep sampling
- Intervention arm 2 (Experimental): Dry one, where FloqSwab, with which perform the sampling is contained and will be preserved after sampling in a tube without preservation solutions
  Interventions: Device: Self sampling device
- Intervention arm 3 (Experimental): Wet one in which, after sampling, the FloqSwab, will be dissolved in preservation solutions.
  Interventions: Device: Self sampling device

INTERVENTIONS:
Device: Self sampling device — The investigators will allocate randomly the women to two different self sampling devices differing in having or not a preservative buffer
  Arms: Intervention arm 2; Intervention arm 3
Other: Cervical ThinPrep sampling — Women are inviated with a standard invitation letter to perform cervical ThinPrep sampling at the clinic on a pre-fixed date
  Arms: Control arm 1

SUMMARY:
The aims of the present study are to assess the effects of a hrHPV self-sampling test as strategies to reach non-attending women in organized cervical screening in comparison with standard recall by letter in 8000 women; to evaluate the performance of two self sampling devices with and without a preservative buffer and to explore their acceptability among invited women and to evaluate a molecular triage approach for management of HPV positive women in self sampling collected material by HPV genotyping and DNA methylation marker panel

DETAILED DESCRIPTION:
The study will be performed in the Tuscany Region including three organised screening programmes : Florence, Viareggio, and Carrara. In these areas, cervical screening programmes actively invite all the resident female population aged 34-64 years for HPV (Human Papilloma Virus) test as primary screening test (Florence and Viareggio), according to the new protocol for cervical cancer screening in Tuscany Region, or Pap-test every 3 years (Carrara). Women aged 34-64 years who had been invited by the screening programme in the previous round of screening and had failed to respond for at least 3 years will be eligible for mail recall.

In the 3 involved screening programs , every year about 63.000 in the age class 34-64 years are invited to participate at the screening program and about 40% of women do not responded to the invitation of the program. Out of them, 8000 eligible women consecutively selected from the lists will be randomised in two groups. The aim is to evaluate the response rate to invitation to a self obtained vaginal-cervical sample for hr-HPV infection testing in comparison to the standard written reminder letter. Randomisation will be performed centrally by the coordinating centre (ISPO) using computer generated random numbers. In the first year a random sample of 4000 eligible women from the 4 screening programs will be invited to participate in the study sending self sampling at home. In the control arm , the women will receive the usual recall with a new invitation letter with a prefixed appointment (it can be moved with a phone call) to perform HPV screening test in the local districts or clinic. In the intervention arm selected to receive self sampling at home, the investigators will allocate randomly the women to 2 different self sampling devices differing in having or not a preservative buffer.

So the group of women allocated in the intervention arm (4000) will be further randomized 1:1 for receiving S-wet or S-dry device .

Assuming that the compliance for the traditional method with an invitation letter is equal to 15% (Giorgi Rossi 2010), the present study is designed to be able to detect an absolute difference of 1.5% or greater in the attendance rate with a conventional levels of power (80%) and significance (95%, one side test) with a planned sample size of 8000 women. Assuming a sample size equal to 2000 women for each sampling devices, a significant difference equal to or greater than 4.0 percentage points more or less , considering a HPV positive rate of about 21% (Giorgi Rossi 2010) with same power and significance.

The study will be submitted , before starting, for approval to the Coordinating Center and Area Vasta Local Ethical Committees. Each women in the study groups will receive an alerting letter explaining that the local Public Screening Program would provide her with a box containing a self-sampler device completely free of charge to perform self- HPV screening test directly at home. After 1 week, each screening program involved in the study will ship by regular mail at home of the randomised women a letter of invitation to participate in the HPV screening program and a box with: self-sample sampling device, a HPV screening leaflet in use in Tuscany Region Program. Information related to the study, instructions to perform self-sampling, pre-printed labels to put on the tube, the informed consent form to sign , the questionnaire and a pre-stamped envelope to return the self-sampling kit. Questionnaires will be send with self-sampling device including items related to: date of women's latest Pap-test, questions about the self-sampling performance (pain, embarrassment, feasibility), what was mostly appreciated in the self-sampling (doing it by themselves, privacy, absence of a doctor, absence of speculum) and what they did not like regarding self-sampling (pain, the device, the instruction ). All information will be collected using 5-point ordinal scales on the general acceptability. Women that decide to participate in the study can send directly by regular mail to the local screening program the pre-stamped envelope with the self-sampling, the questionnaire and the signed informed consent (which will also include the authorization for telephone contact). In second year of study in the city of Florence the investigators will also evaluate the possibility to involve Drugstores in the distribution of self-sampling. In this case 500 randomised women will be invited by letter to perform self sampling for HPV screening test collecting the device in the drugstore. A list of drugstores which agreed to be included in the study will be available in the invitation letter. The impact on compliance and satisfaction of women will be evaluated. All HPV analysis and molecular tests will be performed in Molecular Laboratory of ISPO , the central lab for HPV screening test in Tuscany Region

DNA cobas4800 HPV test:

HPV will be evaluated with the same HPV test used in regular screening: the Cobas 4800 HPV test (Roche Diagnostics) is a qualitative in vitro test that utilizes amplification of target DNA by real-time Polymerase Chain Reaction (PCR) for the detection of 14 high-risk (HR) HPV types in a single analysis. It is a qualitative multiplex assay that provides specific genotyping information for HPV types 16 and 18, while concurrently detecting the other 12 high-risk HPV types (31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68) as a pooled result. ß-globin from cellular input is used as an internal control to assess specimen quality. The test is being performed on the completely automated cobas 4800 System (Roche Diagnostics), according to the manufacturer's instructions; a sample is considered positive according to the specific algorithm of the Cobas system software.

Management of enrolled women HPV negative women will receive at home the results of the screening test and they are re-invited after 5 years according to the HPV screening protocol. All women who resulted in being HPV positive will be contacted by phone to perform colposcopy and a counselling on HPV and cervical cancer risk. If the colposcopy will be positive, a biopsy will be taken, and each women will be followed according to the protocol of HPV screening program in Tuscany. If colposcopy will be negative, women will be re-invited to undergo control with HPV test within a year's time. During colposcopy also a Pap test will be taken to guide the post colposcopic follow-up according to the protocol approved in Tuscan Region. If a woman with hr-HPV did not attend, efforts were made to contact her again by phone and then also by letter.

Molecular Triage of HPV positive women

HPV Genotyping :

Specific genotyping will be performed in all hrHPV positive samples. DNA extracted will be genotyped. In all HPV positive self-collected samples the investigators will perform quantitative methylation analyses in order to obtain a quantification for the methylation status of the investigated CpGs, using DNA extracted for genotyping. The investigators will evaluate Methylation of CpG islands within promoter regions of genes and microRNAs such as CADM1 (Cell adhesion molecule 1), MAL (Myelin and lymphocyte protein), and hsa-miR-124- and methylation status of the HPV regions L1 and L2. The investigators will investigate for each type the CpGs located nearby the sequence position of HPV16 CpGs which have been highlighted as associated with an increased risk of cervical intraepithelial neoplastic (CIN2+) disease: L1 nucleotide positions 5601-5616 and 6457; L2 nucleotide position 4261.

Bisulfite modification: Genomic DNA samples will undergo bisulfite modification using the commercial EpiTect Bisulfite Kit (QIAGEN). The bisulfite-modified genomic DNA will be used immediately for pyrosequencing or stored at -80°C.

Human synthetic methylated and unmethylated DNA controls for human genes and DNA from CaSki cell line or a WHO (World Health Organization) HPV16-DNA control for viral genes will be included in each modification set to check modification efficiency.

Methylation status: Methylation status in the selected genes will be evaluated on the bisulfite modified DNA. The assays will be performed employing primers selected according to published sequences (Hesselink AT et al. Mirabello L et al, Wentzensen N et al). When not available, primers will be designed using a specific software . Links with available Gene-banks will be set up for gene sequence references. A preliminary PCR reaction will be performed in a total volume of 35 microL containing 1X KCl, 2mM MgCl2 , 200 microM dNTPs, 0.5 microM of each primer (antisense biotinylated), 1.75U Taq polymerase and 6 microL modified DNA with the proper thermocycling profile. Amplification and real-time measurement was performed in the 7500 ABI system (Applied Biosystems, Foster City, CA, USA). Bisulfite modified controls for methylated and unmethylated status of cell and viral gene respectively will be included in each run.

Genotyping and Methylation results will be correlated in terms of sensitivity and specificity to histological outcome and follow-up results in HPV positive women with and without clinically meaningful cervical disease diagnosed within a two-year follow-up period.

Role of each Unit involved in the study and timeline In the first year of the study ISPO will select and randomise women , set up the study data base and the software computer validation. The boxes and all materials for the mailing of self sampling devices will be prepared.

Each screening center will invite women, will send the box with self sampling device, receive the self sampling device from the invited women, register them in the database, send the samples to ISPO. ISPO L.R.P.O (Regional Oncological Prevention Laboratory) will perform hr-HPV testing and send the results to each screening center. Each screening center will receive the hr-HPV results from ISPO and send them to the woman. In case of HPV positive results the local screening center will contact the woman by phone for colposcopic assessment, perform colposcopy and every further follow-up visits, record the results and questionnaires data in the data base and participate in evaluation of the results.

In the second year ISPO will evaluate the feasibility to distribute the self sampling using pharmacies and invited women for this purpose performing hr-HPV test for responding women. ISPO will perform also HPV typing and methylation profiles, will records all data in the data base of the study, perform statistical analysis and evaluation of the results.

ELIGIBILITY:
Inclusion Criteria:

Not responding to the previous screening round

Exclusion Criteria:

Had any cervical smears taken for < 3 years

Pregnant

Ages: 34 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8000 (Estimated)
Dates: Start 2016-08-09; Primary Completion 2017-08-09 (Actual); Study Completion 2018-08-09 (Estimated)

PRIMARY OUTCOMES:
hrHPV self-sampling test | 14 months
  Effects of a hrHPV self-sampling test as strategies to reach non-attending women in organized cervical screening

SECONDARY OUTCOMES:
Evaluation of collection and storing performance of two self sampling devices | 14 months
  Will be evaluated the performance of two collection systems in terms of collecting and storing the biological material for consecutive molecular analysis.

OTHER OUTCOMES:
Evaluation of the best triage strategy for self samples | 14 months
  The study provides that all HPV positive women of the active arm of the study will perform colposcopy. On the HPV positive woman samples the investigators carry out the molecular analysis to evaluate various molecular triage strategies (HPV genotyping, methylation of human genes (MAL-1, CADM1, hsa-miR-124-2) and methylation of viral genes L1 and L2). The molecular marker's results will be compared with the colposcopic results to evaluate its sensitivity, and specificity.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca M Carozzi, PhD, Principal Investigator — Cancer prevention and Research Institute
Locations (1):
- Cancer Prevention and Research Institute, ISPO, Florence, FI, Italy

REFERENCES:
- [Background] Giorgi Rossi P, Marsili LM, Camilloni L, Iossa A, Lattanzi A, Sani C, Di Pierro C, Grazzini G, Angeloni C, Capparucci P, Pellegrini A, Schiboni ML, Sperati A, Confortini M, Bellanova C, D'Addetta A, Mania E, Visioli CB, Sereno E, Carozzi F; Self-Sampling Study Working Group. The effect of self-sampled HPV testing on participation to cervical cancer screening in Italy: a randomised controlled trial (ISRCTN96071600). Br J Cancer. 2011 Jan 18;104(2):248-54. doi: 10.1038/sj.bjc.6606040. Epub 2010 Dec 21. PMID 21179038
- [Background] Gok M, Heideman DA, van Kemenade FJ, Berkhof J, Rozendaal L, Spruyt JW, Voorhorst F, Belien JA, Babovic M, Snijders PJ, Meijer CJ. HPV testing on self collected cervicovaginal lavage specimens as screening method for women who do not attend cervical screening: cohort study. BMJ. 2010 Mar 11;340:c1040. doi: 10.1136/bmj.c1040. PMID 20223872
- [Background] Gok M, van Kemenade FJ, Heideman DA, Berkhof J, Rozendaal L, Spruyt JW, Belien JA, Babovic M, Snijders PJ, Meijer CJ. Experience with high-risk human papillomavirus testing on vaginal brush-based self-samples of non-attendees of the cervical screening program. Int J Cancer. 2012 Mar 1;130(5):1128-35. doi: 10.1002/ijc.26128. Epub 2011 May 30. PMID 21484793
- [Background] Hesselink AT, Heideman DA, Steenbergen RD, Coupe VM, Overmeer RM, Rijkaart D, Berkhof J, Meijer CJ, Snijders PJ. Combined promoter methylation analysis of CADM1 and MAL: an objective triage tool for high-risk human papillomavirus DNA-positive women. Clin Cancer Res. 2011 Apr 15;17(8):2459-65. doi: 10.1158/1078-0432.CCR-10-2548. Epub 2011 Mar 9. PMID 21389098
- [Background] Holanda F Jr, Castelo A, Veras TM, de Almeida FM, Lins MZ, Dores GB. Primary screening for cervical cancer through self sampling. Int J Gynaecol Obstet. 2006 Nov;95(2):179-84. doi: 10.1016/j.ijgo.2006.07.012. Epub 2006 Sep 25. PMID 16997304
- [Background] Igidbashian S, Boveri S, Spolti N, Radice D, Sandri MT, Sideri M. Self-collected human papillomavirus testing acceptability: comparison of two self-sampling modalities. J Womens Health (Larchmt). 2011 Mar;20(3):397-402. doi: 10.1089/jwh.2010.2189. Epub 2011 Feb 25. PMID 21351869
- [Background] Khanna N, Mishra SI, Tian G, Tan MT, Arnold S, Lee C, Ramachandran S, Bell L, Baquet CR, Lorincz A. Human papillomavirus detection in self-collected vaginal specimens and matched clinician-collected cervical specimens. Int J Gynecol Cancer. 2007 May-Jun;17(3):615-22. doi: 10.1111/j.1525-1438.2006.00835.x. PMID 17504376
- [Background] Lazcano-Ponce E, Lorincz AT, Cruz-Valdez A, Salmeron J, Uribe P, Velasco-Mondragon E, Nevarez PH, Acosta RD, Hernandez-Avila M. Self-collection of vaginal specimens for human papillomavirus testing in cervical cancer prevention (MARCH): a community-based randomised controlled trial. Lancet. 2011 Nov 26;378(9806):1868-73. doi: 10.1016/S0140-6736(11)61522-5. Epub 2011 Nov 1. PMID 22051739
- See also: Related Info — http://www.ispo.toscana.it